CLINICAL TRIAL: NCT05199935
Title: A Randomized Controlled Trial Comparing the Effectiveness of a Safety-promoting Intervention With Standard Antenatal Care for Pregnant Women in Nepal
Brief Title: Testing the Effectiveness of a Safety-promoting Intervention in Antenatal Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Kathmandu Medical College and Teaching Hospital (Other); Kathmandu University School of Medical Sciences (Other); University of South-Eastern Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 178092
Record Dates: First submitted 2022-01-05; First posted 2022-01-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Domestic Violence
Keywords: Pregnancy; Nepal
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Intervention Model Description: A two armed randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All participants will view a video twice. At baseline (Time 0) one group will view the intervention video and the other group the control video. Both video are of the same length. Women are seated in such a way that they cannot view each others screens. All women will view the intervention video after the main outcome has been collected at time 1. Care providers will provide standard care and not know which group women in unless they specifically ask at which point the woman viewed a video and if she talked to someone in person after viewing the video. The data-set will be masked so that the statistician analyzing will not know the code for the two different groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Are shown the intervention video after filling out baseline questionnaire
  Interventions: Behavioral: Video
- Control (Other): Are shown a control at Time 0, baseline and the intervention video after main outcome data is collected at Time 1
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Video — Information on violence and safety behaviors. Women are encouraged to share their experience of domestic violence with others.
  Arms: Intervention
Other: Control — Control video on healthy pregnancy
  Arms: Control

SUMMARY:
Domestic violence during pregnancy can directly or indirectly cause maternal and fetal morbidity and even mortality. The investigators have validated the Abuse Assessment Screen to the Nepali context for use with a color-coded audio computer assisted self-interview method among pregnant women. This instrument will be used to identify women experiencing domestic violence during or shortly prior to their current pregnancy. In addition, an intervention video was developed. The aim of the video is to encourage women to take safety actions, in particular telling someone about the violence experienced. Women in the control group will watch a video on a healthy pregnancy and sign and symptoms of complications and what to to if these occur.The control video was chosen to increase blinding. This study aims to investigate the effect of the video compared to an intervention video.

DETAILED DESCRIPTION:
This randomized controlled study is a two armed study, which will take place at two locations in Nepal. Eligible women will be invited to the study when attending routine antenatal care. Women agreeing to participate will be invited to first complete a questionnaire. Upon completion of this first questionnaire women will view either the intervention or control video, irrespective of their Domestic Violence (DV) Status. In the intervention arm all women will be shown the intervention video, irrespective of their DV status. In the control arm women view an intervention video. All women are asked to return to the study during the last two months of their pregnancy. All women will be asked to complete the second questionnaire. Upon completions all women will be offered to see the intervention video. For the intervention group this will be their second viewing, for the control group this will be the first viewing of the intervention video. All women will be followed up til birth. Data about their birth will be collected from their hospital records.

ELIGIBILITY:
Inclusion Criteria:

* between 12 to 20 weeks gestational age of pregnancy

Exclusion Criteria:

* prior 12 weeks gestation
* after 20 weeks of pregnancy
* mentally unable to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2230 (Actual)
Dates: Start 2023-01-29 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Seeking support | 12 to 24 weeks after intervention
  A single question asking women if they have told anybody about the experience of domestic violence besides the person at the personal follow-up at Time 1 (baseline)

SECONDARY OUTCOMES:
Ways of Coping Checklist | 12 to 24 weeks after intervention
  Sub-scales seeking social support, avoidance and detachment, self-blame
Use of safety measures | 12 to 24 weeks after intervention
  Measures women can take to prepare for leaving or reduce violence
Change in Domestic Violence status | From baseline (questionnaire nr. 1) to time 1, questionnaire number 2.
  A change in domestic violence status from reporting not any experience of any domestic violence to reporting experience of any domestic violence, or the contrasting result going from reporting the experience of any domestic violence to reporting no experience of any domestic violence.

OTHER OUTCOMES:
Hopkins Symptom Checklist - 10 | 12 to 24 weeks after intervention
  Symptoms of depression and anxiety
Social Acceptance of Wife Abuse Scale | 12 to 24 weeks after intervention
  6 items from the Social Acceptance of Wife Abuse Scale (SAWAS). Minimum score is 0 (zero) and maximum score is 3. A higher score is a worse outcome.
Attitudes towards domestic violence | 12 to 24 weeks after intervention
  WHO set of questions

CONTACTS AND LOCATIONS:
Overall Officials: Schei Berit, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (2):
- Nepal (2):
  - Dhulikhel Hospital, Dhulikhel
  - Kathmandu Medical College, Kathmandu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chalise P, Manandhar P, Infanti JJ, Campbell J, Henriksen L, Joshi SK, Koju R, Pun KD, Rishal P, Simpson MR, Skovlund E, Swahnberg K, Schei B, Lukasse M. Addressing Domestic Violence in Antenatal Care Environments in Nepal (ADVANCE) - study protocol for a randomized controlled trial evaluating a video intervention on domestic violence among pregnant women. BMC Public Health. 2023 Sep 15;23(1):1794. doi: 10.1186/s12889-023-16685-6. PMID 37715147